CLINICAL TRIAL: NCT06785740
Title: StAtins in Frail OldEr Patients with Ischemic Stroke or Transient Ischemic Attack - the Prospective Cohort Study
Acronym: SAFEST-coh
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Prof. dr. Nathalie van der Velde, Professor dr. Nathalie van der Velde, Full Professor Geriatric medicine (internal medicine), Amsterdam UMC, location AMC
Other Study IDs: 2024.0202
Record Dates: First submitted 2024-07-03; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Ischemic Stroke; TIA
MeSH Terms: conditions — Ischemic Stroke | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Rosuvastatin Calcium; Pravastatin; Simvastatin; Fluvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Statin continued: Patients in which the statin was continued after the index event
  Interventions: Drug: Statin
- Statin discontinued: Patients in which the statin was discontinued after the index event

INTERVENTIONS:
Drug: Statin — Statin use
  Other Names: atorvastatin, rosuvastatin, pravastatin, simvastatin, fluvastatin
  Groups: Statin continued

SUMMARY:
Two Dutch guidelines (Stroke and Cardiovascular Risk Management) provide conflicting advice on optimal statin treatment in older patients. In the SAFEST-cohort, the investigators will assess the impact of continuing versus discontinuing a statin in frail individuals aged 70 and above with a recent ischemic stroke or transient ischemic attack (TIA) on their health-related quality of life and MACE free survival during a two-year follow-up period.

DETAILED DESCRIPTION:
The stroke incidence strongly increases with age.Many of the older individuals that suffered a stroke will have to live with stroke sequelae and will need lifelong care, either at home or in a nursing facility.

Hence, secondary prevention strategies are of the highest importance. Statins are used for the prevention of subsequent cardiovascular events in ischemic stroke and TIA patients. The efficacy of statin therapy has been firmly established in middle-aged stroke patients. However, despite the high prevalence of stroke in older people, the evidence for the efficacy of statin therapy in older individuals that suffered an ischemic stroke or TIA is sparse. This primarily arises from the underrepresentation of older patients in statin trials.

In a recent meta-analysis, it was found that in people aged 70 and above, statin use lowered the annual incidence of major vascular events with approximately one percent. However, the trials in this meta-analysis mostly included fit, non-frail older adults.

Frailty is a geriatric condition characterized by an increased vulnerability to external stressors, linked to adverse outcomes, including premature mortality. A considerable proportion of the older population is frail. However, since trials that include older individuals often focus on fit, non-frail older adults, there is currently no evidence for the most effective treatment strategy in the frail older group.

While it might be tempting to extrapolate the benefits of statin therapy from younger patients to frail older patients, it is vital to acknowledge the considerable disparities between these groups. Firstly, frail older stroke survivors may not have a life-expectancy longer than the time to benefit. Secondly, due to the high percentage of polypharmacy in frail older people, this patient group has a higher risk for the occurrence of drug-drug interactions and adverse effects, which have the ability to significantly affect the quality of life.

The limited body of evidence regarding the effectiveness of statins in the older population, combined with their higher susceptibility to side effects and drug interactions, results in uncertainty for patients as well as for doctors and policymakers when deciding how to treat this patient group.This uncertainty is clearly reflected in the two Dutch guidelines ("Herseninfarct en Hersenbloeding" and "Cardiovascular Risk Management (CVRM)" respectively), providing conflicting advice on optimal statin treatment in older patients.

The investigators hypothesize that in frail older patients with a recent ischemic stroke or TIA, discontinuing statins will increase health-related quality of life (HrQoL) without a substantial decrease in Major Adverse Cardiovascular Events (MACE) free survival, which includes cardiovascular death, nonfatal myocardial infarction (MI), or nonfatal stroke.

In this prospective cohort study, no intervention will be implemented. Participants will be followed for two years (and for the patients included in the first years of the inclusion period - three). During this time, data is collected including questionnaires on quality of life, occurrence of MACE or falls, and possible changes in statin treatment.

ELIGIBILITY:
Inclusion Criteria:

* age = 70 years or older at the time of ischemic stroke or TIA;
* inclusion within 6 weeks after diagnosis of ischemic stroke or TIA;
* already using statin therapy at the time of the index event;
* frailty as defined by a pre-event score of 4-7 and/or post-event score of 6-7 on the validated Clinical Frailty Scale.

Exclusion Criteria:

* Previous serious adverse drug reactions (defined as an adverse reaction that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisa-tion, results in persistent or significant disability or incapacity, or is a birth defect32) to statins or other contraindications to statin use.
* Very severe frailty or very limited life expectancy (< 6 months) as defined by a score >= 8 points on the validated Clinical Frailty Scale.
* Inability to communicate in Dutch.
* Inability to respond to questions, either independently or with the assistance of a proxy.
* Inability or unwillingness to provide written informed consent, either independently or with the assistance of a proxy.

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: frail individuals aged 70 and above with a recent ischemic stroke or transient ischemic attack (TIA)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HrQoL) | 3, 6, 12, 18, 24 (and 36) months
  This will be measured using the PROMIS-10 scale scores (ranging from 0 to 100, with higher scores indicating better health), including global mental health and global physical health subscales. Measurements at 3, 6, 12, 18, 24 (and 36) months.
  months.
Major Adverse Cardiovascular Events (MACE) free survival | 3, 6, 12, 18, 24 (and 36) months
  Classical 3-point MACE (cardiovascular death, nonfatal MI, or nonfatal stroke) and non-cardiovascular death.
  Measurements at 3, 6, 12, 18, 24 (and 36) months.

SECONDARY OUTCOMES:
Functional outcome | 3, 6, 12, 18, 24 months
  This will be assessed using the modified Rankin Scale (mRS), with scores ranging from 0 to 6 (lower scores indicating better function).
Cognition | 3, 6, 12, 18, 24 months
  This will be measured using the Montreal Cognitive Assessment (MoCA) with scores ranging from 0 (worst) to 30 (best) or the Telephone version of the MoCA (TMoCA) with scores ranging from 0 (worst) to 22 (best)
Number of falls | 3, 6, 12, 18, 24 months
  Falls, measured using the falls calender. Participant returns the fall calender every 3 months.
Time to first fall | 3, 6, 12, 18, 24 months
  Falls, measured using the falls calender. Participant returns the fall calender every 3 months.
General quality of life using the EQ-5D-5L | 3, 6, 12, 18, 24 months
  General QoL, measured by the EuroQol Questionnaire (EQ-5D-5L), with scores ranging from 0-100, the higher, the better.
Societal costs | 3, 6, 12, 18, 24 months
  Societal costs measured by The Older Persons and Informal Caregivers Survey - Minimum Data Set (TOPICS-MDS) (questions 23 - 37)
Cardiovascular risk status | 3, 6, 12, 18, 24 months
  This will be assessed by collecting vital signs (height, weight, and blood pressure) and lipid levels. The exact way how to combine these factors into one risk status will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Renske van den Berg-Vos, Prof. dr., Principal Investigator — Amsterdam UMC, Academic Medical Center, University of Amsterdam, Amsterdam, The Netherlands; Nathalie van der Velde, Prof. dr., Principal Investigator — Amsterdam UMC, Academic Medical Center, University of Amsterdam, Amsterdam, The Netherlands
Locations (4):
- Netherlands (4):
  - Flevoziekenhuis, Almere Stad
  - Amsterdam UMC, location AMC, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
The SAFEST database can be requested by other researchers. These requests will be reviewed according the requirements for sharing SAFEST data.
Supporting Information: Study Protocol, SAP
Time Frame: After data-collection/analysis.
Access Criteria: Requirements for sharing SAFEST data include:
  * privacy laws of the Netherlands, policy of NFU and AmsterdamUMC must be followed
  * data will be anonymously shared
  * data can only be used to study the research question for which participants signed the ICF
  * data will not be shared for commercial purposes.